CLINICAL TRIAL: NCT05109806
Title: Psychological Functioning of Children & Adolescent With Congenital Heart Disease, and Their Parents: An Intervention Based Study
Brief Title: Psychological Functioning of Children and Adolescents With CHD andTheir Parents, An Intervention Based Study
Acronym: CHDPIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Asma Riaz Hamdani, Lecturer, Government College University Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHDPIM1981
Record Dates: First submitted 2021-09-04; First posted 2021-11-05 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Congenital Heart Disease; Psychological Intervention; Parenting; Quality of Life; Psychological Disturbance
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: The study has already approved from FIC a tertiary care unit for ethical committee review. Personal informed consent of patients and their parents will also be taken. Before starting the phases of study all the permissions regarding the measures will also be taken from original authors.
  The registered participant in 1st study will get information letters explaining the purpose and the content of the study. All the participants will be given a research card and reference code for registration and information. Randomization: After informed consent have been obtained, Families will receive an anonymous study code and will be invited for medical and psychological baseline assessments. Thereafter, All participants will be randomly assigned to experimental and control groups.
Who Masked: Participant
Masking Description: participants are only blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Problem prevention therapy will be given as per intervention. a group of parents will be included for a group session for narration of their problems in relevance to health related quality of life .After the assessment the next session the solution to these problems would be given to them.
  Interventions: Behavioral: problem prevention therapy with CHD
- control group (Other): for this group only a general education regarding disease will be conducted and no further interventions will be provide to them .
  Interventions: Behavioral: problem prevention therapy with CHD

INTERVENTIONS:
Behavioral: problem prevention therapy with CHD — The psychological exercises are based on the evidence-based Fun FRIENDS protocol (Burhanar, 2016) for reducing emotional behavioral issues. Separate workshop of adolescents will be designed based on transition in child cardiology to adult cardiology(Moons et al., 2009) . A cardiologist and psychologist will psycho educate them about self-care, needs of transition period and strength and strains about further life.
  Other Names: psycho education

SUMMARY:
Almost 1% of infants are born with Congenital Heart Disease (CHD), an umbrella term referring to a range of anomalies in the heart's structure that are present at birth. Owing to significant medical advances, it is now estimated that more than 90% of persons born with CHD will reach adulthood. Children with CHD and their families' mental health outcomes need for psychosocial care. This study will intend to improve the psychological functioning of children, adolescents with CHD and their parents. The research will comprise of two major studies. The sample of first study will be based on a Cohort (From April 2021 to October 2021) of children, adolescent and their parents. Participants will be assessed for their psychological functioning and health related quality of life using Strength and Difficulty Questionnaire, pedsQL 3.0 cardiac module , Parental Stress Index , and 36-Item Short Form Survey. It is hypothesized that parental psychological functioning will mediate the relationship between psychological functioning of children and adolescent with CHD and their health related quality of life. It is also hypothesized that emotional behavioral issues of children and adolescents will moderate the link between parental psychological functioning and their quality of life. Illness parameters and sociodemographic correlates will serve as covariates in the study. This study will provide a baseline for the second study that is expected to use a randomized control trial of an intervention program based on training workshops derived from CHIP for the reduction in parental distress, emotional behavioral problem and improvement in health related quality of life among children, adolescent with CHD and their parents. The pretest-posttest design will be used. The randomized control trial will be conducted as per Consort Guidelines. A sub sample will be selected from the initial study using purposive sampling. Intervention study will include a subsample of CHD population (60 children and adolescents each) and their parents using purposive sampling technique. The participants will be randomly assigned to experimental & control groups. Illness related and demographic parameters will be distributed equally in both groups for establishing control. The intervention will be administered to experimental group only, while control group will receive regular treatment. Results of Pretest and posttest measures will be statistically analyzed. The designed intervention program (using problem solving therapy, psycho-education and Parenting the child with CHD training) will lower the level of parental stress in parents and emotional behavioral issues in CHD population. It will further increase the level of health related quality of life among children and adolescent with CHD and their parents. The research will incorporate psychosocial care with CHD population along with their regular treatment and thus improve their future health related outcomes in Pakistan.

DETAILED DESCRIPTION:
The approved clinical trial is a part of PhD research project entitled as ,"Psychological Functioning of Children and Adolescents with congenital Heart Disease, and Their Parents: An Intervention based study ". The study aims to assess the psychological functioning of CHD population in early years of life and evaluating its outcomes on their parents psychological health. Furthermore the clinical trials have designed to check the efficacy and utility of an Intervention Program for improving the quality of parenting and health related quality of life in children and adolescent with congenital heart disease.

The Randomized Control Trials will be used to check the utility of this intervention program. The intervention is derived from CHIP school, CHIP family and psychological intervention for CHD patients Design A two arm cluster controlled trial will be carried out at Pediatric Cardiology Department, FIC. This work will be conduct with the collaboration of a paeds cardiologist from FIC and their staff.

Participants All the participants who had registered and given consent in 1st study (From April 2021 to October 2021) will serve as the target population for the 2nd study. Families from the study one will be provided with the information about the second study and consent will be sought again for participation in this study. A purposive sample (n=60) of children adolescent and their families will be taken as participants in this study.

Inclusion Exclusion Criteria Parents of children with CHD below age 10 will be enrolled for the RCT trial. A sub sample considering the psychological portfolio obtained from the 1st study using purposive sampling technique will be recruited for both experimental and control group. Children with comorbidities and neurological deficits will be excluded.

Ethical Consideration The single blinded parallel randomized controlled trial has been approved by of Ethical Review Board of Faisalabad Institute of Cardiology (FIC) and University Ethical Committee of Government college university, Faisalabad. The registered sample will be informed about the nature and the purpose of the study. They will have right to choose/quit the study at any time. Informed consent will be obtained from the parents of children and adolescent. Assent from participants above age12 will also be obtained. The trial will be registered at provincial and national trial committee in Pakistan.

Procedure The study has already been approved from the Advanced Studies and Research Board of GC University Faisalabad and Faisalabad Institute of Cardiology, a tertiary care unit for ethical committee review. Personal informed consent of patients and their parents will be taken. Initially, permissions to use the psychological assessment tools will also sought from the original authors.

The registered participant in 1st study will get information letters explaining the purpose and the content of the study. The entire sample will be provided with a research card and reference code for registration and information. Randomization: After obtaining informed consent, families will receive an anonymous study code and will be invited for medical and psychological baseline assessments. Thereafter, controlling for age, gender, and severity of illness, the participants will be randomly assigned into groups (experimental, control).

IMPLICATIONS OF THE STUDY

Following are the implications of the study:

1. The result will establish the efficacy of intervention based psychosocial care of youth with CHD and their parents in Pakistan
2. The research will incorporate psychosocial care with CHD population along with their regular treatment and thus improve their future health related outcomes.
3. The result of the research will facilitate the participating children and adolescents in their transition to adulthood thus helping them to become a functional part of the society.
4. The research outcomes will pave the way for recruitment of health psychologist in pediatric cardiology units in Pakistan.
5. The research will not only help parents to understand disease related physical but also psychological outcomes and facilitate them in managing their own stress and relation with the child according to his psychosocial needs

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents who will be diagnosed with Cyanotic CHD
* able to understand Urdu language
* patient with both gender will be included
* intact families will be included

Exclusion Criteria:

* single parents
* parents having any psychiatric illness
* Any chromosomal abnormality

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Paediatric quality of life | 6month
  The Child and Parent reports of the paedsQl genric core scales for Young Children( ages 5-7) Children(8-12) Teens (13-18) 5 point Likert scale from 0 to 4 .Total scores will be Used to measure Health Related Quality of Life. High score indicate better quality of life .
parenting stress Scale | 6month
  The PSS is an eighteen item questionnaire assessing parent feeling about their parenting role, emotional and positive emotions , personal development and aspects of demands of parent hood. The parent stress scale was developed by Judy Berry and warren jones and can be used to assess outcomes of intervention designed to support parenting efficacy. High scores denotes higher level of stress in parents.

SECONDARY OUTCOMES:
36 item short form survey | 1 year
  The RAND 36 item health survey taps eight concept; physical functioning, Bodily pain, role limitations due to physical health problems and role limitations due to emotional health problems, Energy fatigue and general health. scoring involves two step process first preceded numeric values in second same was average together to create the scale scores. Higher score denotes better general health and well being

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rabia Khawar, PhD, Study Chair — Department of Applied Psychology, GC University Faisalabad; Asma Riaz Hamdani, PhD Scholar, Principal Investigator — Department of Applied Psychology, GC University Faisalabad
Locations (1):
- Government College university ,Faisalabad and Faisalabad Institute of cardiology, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Mheen M, van Beynum IM, Dulfer K, van der Ende J, van Galen E, Duvekot J, Rots LE, van den Adel TPL, Bogers AJJC, McCusker CG, Casey FA, Helbing WA, Utens EMWJ. The CHIP-Family study to improve the psychosocial wellbeing of young children with congenital heart disease and their families: design of a randomized controlled trial. BMC Pediatr. 2018 Jul 12;18(1):230. doi: 10.1186/s12887-018-1183-y. PMID 30001701
- [Background] Lawoko S, Soares JJ. Psychosocial morbidity among parents of children with congenital heart disease: a prospective longitudinal study. Heart Lung. 2006 Sep-Oct;35(5):301-14. doi: 10.1016/j.hrtlng.2006.01.004. PMID 16963362
- [Background] Lisanti AJ. Parental stress and resilience in CHD: a new frontier for health disparities research. Cardiol Young. 2018 Sep;28(9):1142-1150. doi: 10.1017/S1047951118000963. Epub 2018 Jul 11. PMID 29991369
- [Background] Moons P, Pinxten S, Dedroog D, Van Deyk K, Gewillig M, Hilderson D, Budts W. Expectations and experiences of adolescents with congenital heart disease on being transferred from pediatric cardiology to an adult congenital heart disease program. J Adolesc Health. 2009 Apr;44(4):316-22. doi: 10.1016/j.jadohealth.2008.11.007. Epub 2009 Feb 12. PMID 19306789
- [Background] Ogundele MO. Behavioural and emotional disorders in childhood: A brief overview for paediatricians. World J Clin Pediatr. 2018 Feb 8;7(1):9-26. doi: 10.5409/wjcp.v7.i1.9. eCollection 2018 Feb 8. PMID 29456928
- [Background] Samad L, Hollis C, Prince M, Goodman R. Child and adolescent psychopathology in a developing country: testing the validity of the strengths and difficulties questionnaire (Urdu version). Int J Methods Psychiatr Res. 2005;14(3):158-66. doi: 10.1002/mpr.3. PMID 16389892
- [Background] Biber S, Andonian C, Beckmann J, Ewert P, Freilinger S, Nagdyman N, Kaemmerer H, Oberhoffer R, Pieper L, Neidenbach RC. Current research status on the psychological situation of parents of children with congenital heart disease. Cardiovasc Diagn Ther. 2019 Oct;9(Suppl 2):S369-S376. doi: 10.21037/cdt.2019.07.07. PMID 31737543